CLINICAL TRIAL: NCT06426888
Title: Comparison of Scapular Stabilization Exercises and Scapular Mobilizations in Patients With Sub Acromial Pain Syndrome
Brief Title: Comparison of Scapular Stabilization and Mobilizations in Sub Acromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSPT/01723 Gulban Aslam
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Scapular stabilization exercises; Range of motion; scapular mobilization
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental interventional group 1(scapular stabilization exercise therapy) (Experimental): 1. Ball stabilization exercise, 2.Wall push up 3. Wall push up Patients will be treated 3 times per week for 4 consecutive weeks
  Interventions: Other: Experimental interventional group 1(scapular stabilization exercise therapy)
- Experimental :interventional group II (scapular mobilizations) (Experimental): scapular mobilization in elevation, depression, protraction and retraction. Patients will be treated 3 times per week for 4 consecutive weeks
  Interventions: Other: Experimental :interventional group II (scapular mobilizations)

INTERVENTIONS:
Other: Experimental interventional group 1(scapular stabilization exercise therapy) — Ball stabilization exercise: While standing close to the wall, the participant will be asked to position her affected hand on the ball and keep the ball from moving as disturbance will be applied in different directions.
  Wall push up: While facing wall patient will be asked to place both hands on wall, shoulder width apart. He will be instruct to breath in, bend his elbows, lean into wall and hold this position for one second then breath out slowly push back until arms are straight again Wall slides
  • Patient will be asked to lean his head, upper thorax and butts against the wall, place his hands and arms against the wall in high five position.
  Arms: Experimental interventional group 1(scapular stabilization exercise therapy)
Other: Experimental :interventional group II (scapular mobilizations) — Patient lies on unaffected side close to the edge of the treatment bench with hips and knees bent for stability.
  Therapist will start by supporting the patient arm on his/her forearm so that shoulder is in maximally loose pack position.
  Then he/she will grab on the scapula with both hands. One hand supports the scapula from cranial around the acromion and scapular spine and other hand from the caudal at the inferior angle of scapula.
  Then both hands move the scapula cranially over the thorax into elevation and caudally into the depression, upward/downward rotation as well as retraction and protraction.
  Arms: Experimental :interventional group II (scapular mobilizations)

SUMMARY:
The aim of this research is to compare the effect Comparison of scapular stabilization exercises and scapular mobilizations on shoulder pain, scapular kinematics, disability and functional limitations in patients with sub acromial pain syndrome Randomized controlled trials done at District Head Quarters Mirpur AJK. The sample size was 36. The subjects were divided in two groups, 18 subjects in scapular mobilization exercise group and 18 in scapular mobilization exercise therapy group. Study duration was of 12 months. Sampling technique applied was non probability convenient sampling technique. Only 25-40 years old patient with unilateral shoulder pain lasting >6 weeks were included. Tools used in the study are NPRS, SPADI, WORC LSST and SAT.

DETAILED DESCRIPTION:
Sub acromial pain syndrome (SAPS), an up to date terminology (shoulder impingement syndrome ) is a common healthcare problem, especially in adult where the space directly below the acromion process and above the shoulder joint, has narrowed and patients describe pain on lateral and anterior aspect of shoulder . The estimated prevalence in the general population is 7 to 26 percent and it accounts for 44 to 65% of all shoulder problems. Incidence of shoulder impingement in the US military population is 7.77 cases/1000 person-years and in UK 3 out of every 4 patient with shoulder pathologies are seeking medical treatment for SAPS. Risk factors include repetitive activity above the shoulder, decubitus sleeping position, a hook-type acromion, smoking, muscle imbalance, bone and joint abnormalities etc. Common symptoms are persistent pain without any history of trauma, difficulty reaching up behind the back, weakness in shoulder muscles, pain when the arm is raised between 70 and 120 degrees and scapular dyskinesia.

* Research surrounding sub acromial pain syndrome has experienced significant growth recently especially in the area of its management. Physiotherapy management protocol for SAPS includes, postural correction exercises, neuromuscular control exercises, Stretching's, manual therapy techniques of the shoulder, scapular stabilization and Mobility Exercises and myofacial release therapy. Scapular stabilization exercises based on open and closed kinetic chain exercises to increase muscle strength and joint position awareness.

ELIGIBILITY:
Inclusion Criteria:

* ● Unilateral shoulder pain lasting >6 weeks

  * Patients with 3/5 positive special tests (Hawkins-Kennedy test, painful arc test, Neer test, Job test, resisted external rotation test)
  * Patients score falling above 3 on NPRS

Exclusion Criteria:

* • History of surgery, fracture, or dislocation in past 6 months

  * Traumatic onset of pain.
  * received steroid injections and physical therapy during the previous 6 months
  * BMI above 30

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | baseline to 4 weeks
  It has 21 items, exploring 5 different domains: Physical symptoms, Sports and recreation, Work, Social function, Emotions. Each question uses a visual analogue scale (VAS) - which is a straight line, representing a 100-point scale, ranging from 0-100.
Lateral Scapular Slide Test (LSST) | baseline to 4 weeks
  this test measures the distance between inferior angle of scapula and nearest vertebral spinous process using tape or goniometer in neutral, 45 and 90 degrees of shoulder abduction with the arms fully internally rotated

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | baseline to 4 weeks
  SPADI measures pain and disability related to shoulder pain and It has 13 items with response options ranging from 0(no pain) to 10 (worst pain), the overall score ranges from 0 to 100.
Numeric pain rating scale | baseline to 4 weeks
  This is an 11 point outcome measure used to measure intensity of pain ranging from 0 (no pain) to 10 (worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- District Head Quarters, Mirpur, Azad Jammu Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No